CLINICAL TRIAL: NCT03400215
Title: Gradient-Echo Spectroscopic Imaging Study of Saturated Fat and Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-01549
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Breast cancer confirmed by biopsy (Active Comparator): Cases will be women first diagnosed with invasive breast cancer confirmed by biopsy
  Interventions: Diagnostic Test: Diagnostic Breast Cancer Scan; Diagnostic Test: Research Scan for Gradient-echo Spectroscopic Imaging (GSI)
- Women without any history of breast cancer (Active Comparator): No known malignancy confirmed by at least 1-year follow up exams.
  Interventions: Diagnostic Test: Diagnostic Breast Cancer Scan; Diagnostic Test: Research Scan for Gradient-echo Spectroscopic Imaging (GSI)

INTERVENTIONS:
Diagnostic Test: Diagnostic Breast Cancer Scan — clinically indicated diagnostic breast MRI scans
Diagnostic Test: Research Scan for Gradient-echo Spectroscopic Imaging (GSI) — 15-min research MRI scan
  Other Names: Gradient-echo Spectroscopic Imaging

SUMMARY:
The role of fat in breast cancer development and growth has been studied extensively using body mass index, a measure of whole body fatness, and dietary fat intake in a number of epidemiological studies. However, there is a paucity of studies, on an individual level, to assess the role of breast fat itself in breast cancer due to lack of a non-invasive and fast measurement method. Since breast fibroglandular cells are surrounded by breast fat cells, the characteristics of breast fat may have a stronger relationship with breast cancer development, as supported by recent studies showing that a majority of breast cancer develops at the interface between fibroglandular tissue and adipose tissue. However, it is not trivial to study the role of breast fat, mainly due to the lack of a non-invasive and fast measurement method sensitive enough to important features of breast fat, such as types of fat.Recently, we have developed a rapid MRI method, referred to as Gradient-echo Spectroscopic Imaging (GSI), to measure fatty acid composition during clinical breast MRI exams. GSI can provide map of saturated fat and unsaturated fats in the breast adipose tissue without performing tissue biopsy. Our pilot study found that the postmenopausal women with aggressive breast cancer, known as invasive ductal carcinoma, have a significantly higher percentage of saturated fat in their breast adipose tissue than the postmenopausal women with only benign lesions.

DETAILED DESCRIPTION:
The overarching goal of this study is to determine the role of saturated fatty acid in breast cancer development and growth. In this proposal, GSI will be used for non-invasive in vivo measurement of saturated fat in the breast adipose tissue of postmenopausal women who undergo diagnostic breast MRI exams (Aims 1 and 2) or MRI-guided biopsy scans (Aim 3). The central hypotheses is that (i) the breast saturated fatty acid fraction measured by GSI is associated with the presence of malignant lesions in the breast and (ii) the breast saturated fatty acid fraction correlates positively with inflammation in the breast adipose tissue that may lead to increase in estrogen production in adipocytes.The proposed study will evaluate whether breast saturated fat is an independent risk factor for breast cancer, and whether it can provide additional diagnostic information to current clinical diagnostic exams. In addition, the proposed imaging measure of breast saturated fat can be used to assess the efficacy of any intervention to reduce cancer-related inflammation in the breast adipose tissue and to investigate the possible role of fatty acid composition in prevention and clinical management of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to MRI scanning (pacemaker, implanted metallic objects, severe obesity or other condition that leads to difficulty lying in the magnet)
* No contraindication to gadolinium contrast agent (severe renal insufficiency (EGFR<30), allergy to gadolinium) which will be injected for clinical exam
* Able and willing to provide informed consent
* Post-menopausal age > 25 years.

Exclusion Criteria:

* Contra-indication to MRI or gadolinium contrast agent (have a pacemaker, aneurysm clip, or other metallic implant; weigh >135 kg; or have renal impairment)
* Breast surgery within prior 12 months, or breast implants
* Any hormonal therapy

Ages: 25 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 135 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
To compare GSI-measured breast SFA fraction between women with malignant and benign lesions. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Linda Moy, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States